CLINICAL TRIAL: NCT05802784
Title: Hysteroscopic Septoplasty by Different Modalities: A Randomized Clinical Trial
Brief Title: Hysteroscopic Septoplasty by Different Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Moustafa Alsayed Alamely, Assistant lecturer of Obstetrics and Gynecology, Mansoura University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD.20.05.324
Record Dates: First submitted 2023-03-22; First posted 2023-04-07 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Septate Uterus; Recurrent Pregnancy Loss; Subfertility
MeSH Terms: conditions — Septate Uterus; Infertility

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scissors arm (Active Comparator): Patients in this group had undergone resection of the septum with hysteroscope and scissors, The scissors used was pointed, single action and semi rigid . Saline was used as the distending medium in the scissors group. Septal incision was carried out using shortening technique by incising the septum at the leading edge and continue dividing by moving from side to side (in narrow septum), or by thinning technique by which incisions will be made along each side of the septum alternately from one cornual end to the other (in broad septum). The operation was stopped if the fluid deficit exceeded 2500 ml of saline.
  Interventions: Procedure: Hysteroscopic septoplasty with scissors
- Resectoscope arm (Active Comparator): Patients in this group had undergone resection of the septum with Monopolar 26 French resectoscope Dilation of cervical os with Hegar's dilator (up to hegar 8 or 9) , incision of the septum using a resectoscope with the Collins knife, monopolar energy (cut 40-70 Watt) and glycine 1.5% as the distension medium, using shortening or thinning incision. The operation was stopped if the fluid deficit exceeded 1000 ml of glycine. The delivery of distension media was conducted by automated pressure delivery system. All patients were prescribed cyclic estrogen and progesterone for two months.
  Interventions: Procedure: Hysteroscopic septoplasty with resectoscope

INTERVENTIONS:
Procedure: Hysteroscopic septoplasty with scissors — In hysteroscopic septoplasty with scissors arm, incision of the septum was done by continuous flow hysteroscopy and scissors using saline as distension media.
  Arms: Scissors arm
Procedure: Hysteroscopic septoplasty with resectoscope — In hysteroscopic septoplasty with resectoscope arm, incision of the septum was done by 26 Fr monopolar resectoscope with collin's knife using glycine1.5% as distension media.
  Arms: Resectoscope arm

SUMMARY:
The goal of this clinical trial is to compare in participant population ( women with uterine septum meeting the inclusion criteria) hysteroscopic septoplasty by resectoscope compared to hysteroscopic septoplasty with scissors.

The main questions to answer are:

Is there a difference in operative time ? Is there a difference in fluid used and fluid deficit? Is there a difference in complications? Is there a difference in reproductive outcome? Researchers will compare the 2 different techniques to see if there is any difference in operative outcome ( operative time, fluid used and deficit, need for second intervention, and operative and postoperative complications) and reproductive outcome.

DETAILED DESCRIPTION:
Study design:

Prospective randomized clinical trial

Study duration and location:

For at least 24 months, Patients admitted to Obstetrics and Gynecology department at Mansoura University Hospital.

Study method

At baseline, the following will be done:

1. History taking: personal history, menstrual history, obstetrical and gynecological history, present and past history.
2. Patient presentation (subfertility or pregnancy loss)
3. Physical examination: General, abdominal and local examination.
4. Diagnosis of uterine septum either by hysterosalpingogram (HSG), Three dimensional transvaginal ultrasound or office hysteroscopy.

Thereafter:

Patients will be prospectively recruited and randomized by computer program to 2 groups

Group A:

Patients in this group will undergo resection of the septum with hysteroscope and scissors. Saline will be used as a distending medium in the scissors group. Septal incision will be carried out using a thinning technique by which incisions will be made along each side of the septum alternately from one cornual end to the other

Group B:

Patients in this group will undergo resection of the septum with monopolar resectoscope , dilation of cervical os with Hegar's dilators , incision of the septum using a resectoscope with the Collins knife, monopolar energy (cut 50-70 Watt) and glycine 1.5% as the distension medium Sample size calculation Sample size was calculated using Power Analysis and Sample Size software program (PASS) version 15.0.5 for windows (2017) using the results published before with the operative duration of hysteroscopic incision in septate uterus by scissors compared to resectoscope as the primary outcome. The study reported the median operative duration as 10 minutes for resectoscope while that for scissors was 30 minutes. The null hypothesis was considered as the absence of difference between both groups regarding the operative duration. A sample size of 16 patients in each group is needed to achieve 95% power (1-β or the probability of rejecting the null hypothesis when it is false) in the proposed study using a two-sided Fisher exact test with a significance level (α or the probability of rejecting the null hypothesis when it is true) of 5% and hypothesized common standard deviation 15 in both groups. 4 patients drop-out is expected, so a total of 20 patients will be enrolled to each group

Statistical analysis Data will be analyzed using the Statistical Package of Social Science (SPSS) program for Windows (Standard version 24). The normality of data will be first tested with one-sample Kolmogorov-Smirnov test.

Qualitative data will be described using number and percent. Continuous variables will be presented as mean ± standard deviation for normally distributed data and median (IQR) for non-normal data. The following tests will be used; Chi square test: Compare qualitative variables. Fisher exact test and monte carlo test: Compare qualitative variables when expected count less than 5.

Independent t- test: Compare two quantitative variables (parametric). Mann Whitney test: Compare two quantitative variables (Non parametric). For all above mentioned statistical tests , the threshold of significance is fixed at 5% level.The results was considered significant when p ≤ 0.05. The smaller the p-value obtained, the more significant are the results.

Ethical consideration:

* Study protocol was submitted for approval by Institutional Review Board
* Approval of the managers of the health care facilities in which the study was conducted.
* Informed written consent will be obtained from each participant sharing in the study.
* Confidentiality and personal privacy will be respected in all levels of the study.
* Collected data will not be used for any other purpose.

ELIGIBILITY:
Inclusion Criteria:

1. Women of reproductive age
2. Seeking conception
3. Diagnosis of a septate or subseptate uterus
4. A history of one of the following:

   * Recurrent pregnancy loss
   * Subfertility
   * Preterm Birth

Exclusion Criteria:

1. Not seeking conception
2. Diagnosis of septate or subseptate uterus with no history of any of the following:

   * Recurrent pregnancy loss
   * Subfertility
   * Preterm Birth
3. Contraindications for surgery
4. Those who refused to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Operative time | During surgery
Fluid deficit | During surgery
Operative and post operative complications | 3 months follow up after intervention
Need for second intervention | 3 months follow up after intervention

SECONDARY OUTCOMES:
Pregnancy rate | At least 6 months follow up after intervention
Live birth rate | Follow up until the end of first clinical pregnancy or 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided